CLINICAL TRIAL: NCT06633861
Title: Data Collection Study for RFP (Respiration From Plethysmogram)
Acronym: SAT+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Collaborators: Betsi Cadwaladr University Health Board (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 200088
Record Dates: First submitted 2024-08-23; First posted 2024-10-09 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: In-patients Assessment of Vital Signs
Keywords: vital signs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- In-patients with routine spot-check monitoring of vital signs (Experimental): In-patients with routine spot-check monitoring of vital signs
  Interventions: Device: spot-check measurement

INTERVENTIONS:
Device: spot-check measurement — Spot-check measurement: different Philips SpO2 sensors and Philips FAST pulse oximeter system, capnography

SUMMARY:
The study will be conducted in hospitalised patients who undergo spot-check monitoring of vital signs as part of their routine care.

DETAILED DESCRIPTION:
In an additional spot-check measurement procedure, the study will measure oxygen saturations through different Philips SpO2 finger sensors. Patients will wear a nasal cannula linked to a CO2 measuring device at the same time. The data from both devices will be used to design and improve algorithms for measurement of respiratory rate with the saturation probe and the Philips FAST pulse oximeter system. The study will include 50 adult patients and 25 pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (aged 18 years or older) willing and able to understand and provide written informed consent
* Paediatric subjects aged 16 years and older willing and able to understand and provide written informed consent
* Paediatric subjects aged approx. 4-16 years and their legal guardians, willing and able to understand and provide written informed consent/assent
* Subject weight within intended use of at least one SpO2 sensor under test at time of enrolment (M1191T: adult patients >50kg, M1196T: adult patients >40kg, M1192A: paediatric patients 15-50kg)
* Willing and able to wear study devices during study procedures
* Subject undergoing regular spot-check measurements as per the site's standard of care

Exclusion Criteria:

* Palliative patients
* Critically ill patients with severe physiological instability (NEWS ≥9)
* Injury/wounds or physical malformation of sensor application site (i.e. fingers, toes, hands, feet)
* Subjects with severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors (self-reported)
* Unwillingness or inability to remove coloured nail polish or artificial nails from application site
* Nail fungus on application site
* Severe dermatitis or hyperkeratosis (e.g. ichthyosis) at sensor application site

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Data collection for database for algorithm development | 6 months
  Anonymized database of subject data from the Oxygen Saturation finger sensors (photoplethysmogram waveform) and the reference sensors (capnography waveform)

CONTACTS AND LOCATIONS:
Overall Officials: Christian P Subbe, Dr., Principal Investigator — Betsi Cadwaladr University Local Health Board
Locations (1):
- Ysbyty Gwynedd Hospital, Wales, Bangor, United Kingdom

IPD SHARING:
Plan to Share IPD: No